CLINICAL TRIAL: NCT05509816
Title: The Effect of Repeat Dosing of Imlunestrant on CYP3A Activity in Healthy Women of Non-childbearing Potential
Brief Title: A Study of Imlunestrant (LY3484356) in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18416; J2J-MC-JZLK (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Imlunestrant

STUDY DESIGN:
Intervention Model Description: This is a fixed sequence, crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam + Imlunestrant (Experimental): Participants received 400 milligram (mg) Imlunestrant (2 × 200 mg) tablets administered once daily (QD) orally for 7 days on Days 3 to 9 and a single dose of 0.5 mg midazolam solution orally on Day 1 and Day 9 as per below dosing sequence:
  Day 1: 0.5 mg midazolam alone Days 3 to 8: 400 mg imlunestrant QD alone Day 9: 0.5 mg midazolam + 400 mg imlunestrant There was a washout period of 8 days between doses of midazolam.
  Interventions: Drug: Midazolam; Drug: Imlunestrant

INTERVENTIONS:
Drug: Midazolam — Administered orally.
Drug: Imlunestrant — Administered orally.
  Other Names: LY3484356

SUMMARY:
The main purpose of this study is to evaluate the effect of imlunestrant (LY3484356) when administered orally on the levels of midazolam in the blood stream in healthy women of non-childbearing potential. The study will also evaluate the safety and tolerability of imlunestrant in healthy women of non-childbearing potential. This study will last up to approximately 6 weeks for each participant including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Women not of childbearing potential
* Participants who are overtly healthy as determined by medical assessment
* Participants with body mass index (BMI) of 18.0 and 35.0 kilograms per meter squared (kg/m²), inclusive

Exclusion Criteria:

* Have known allergies to imlunestrant, related compounds or any components of the formulation or midazolam
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* Use or intend to use medications that are substrate drugs of P-glycoprotein

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - LabCorp CRU, Inc., Daytona Beach, Florida
  - LabCorp CRU, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam + Imlunestrant
Started | 20
Received at Least One Dose of Study Drug | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Midazolam + Imlunestrant: Participants received 400 mg Imlunestrant (2 × 200 mg) tablets administered QD orally for 7 days on Days 3 to 9 and a single 0.5 mg midazolam solution orally on Day 1 and Day 9 as per below dosing sequence:
  Day 1: 0.5 mg midazolam alone
  Days 3 to 8: 400 mg imlunestrant QD alone
  Day 9: 0.5 mg midazolam + 400 mg imlunestrant
  There was a washout period of 8 days between doses of midazolam.
Arm/Group | Midazolam + Imlunestrant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Midazolam
Description: PK: AUC[0-∞] of Midazolam
Time Frame: Day 1: Predose, 0.25hours (h), 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose; Day 9: Predose, 0.25h, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24, 36, 48h postdose
Population: All participants who received at least one dose of study drug (midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 0.5 mg Midazolam: Participants received single dose of 0.5 mg midazolam solution orally on Day 1.
- 0.5 mg Midazolam + 400 mg Imlunestrant: Participants received 0.5 mg midazolam solution orally in combination with 400 mg Imlunestrant (2 × 200 mg) tablets administered orally on Day 9.
Arm/Group | 0.5 mg Midazolam | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20 | 20
nanogram*hour per milliliter (ng*hr/mL) | 12.3 (32) | 11.4 (41)
Statistical Analysis 1: Comparison: 0.5 mg Midazolam vs 0.5 mg Midazolam + 400 mg Imlunestrant; A mixed effects model was used to estimate drug-drug interaction using the Model: Log(PK) = Treatment + Participant + Random Error, where Participant is fitted as a random effect; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric least squares mean = 0.929, 90% CI 2-sided [0.849 to 1.02] — The least square means (LSMs) and differences in LSMs were back transformed to produce the geometric least square means (GLSMs) and ratio between GLSMs. These were reported along with the 90% confidence interval (CI) for the ratio

2. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Midazolam
Description: PK: Cmax of Midazolam
Time Frame: Day 1: Predose, 0.25h, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose; Day 9: Predose, 0.25h, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24, 36, 48h postdose
Population: All participants who received at least one dose of study drug (midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.5 mg Midazolam | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20 | 20
nanograms per milliliter (ng/mL) | 3.84 (35) | 4.12 (31)
Statistical Analysis 1: Comparison: 0.5 mg Midazolam vs 0.5 mg Midazolam + 400 mg Imlunestrant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric least squares mean = 1.07, 90% CI 2-sided [0.989 to 1.16] — The LSMs and differences in LSMs were back transformed to produce the GLSMs and ratio between GLSMs. These were reported along with the 90% CI for the ratio

3. Secondary Outcome: PK: AUC[0-∞] of 1'-Hydroxymidazolam
Description: PK: AUC[0-∞] of 1'-hydroxymidazolam
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug (midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 0.5 mg Midazolam | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20 | 20
ng*hr/mL | 2.75 (40) | 2.26 (40)
Statistical Analysis 1: Comparison: 0.5 mg Midazolam vs 0.5 mg Midazolam + 400 mg Imlunestrant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric least squares mean = 0.821, 90% CI 2-sided [0.777 to 0.868]

4. Secondary Outcome: PK: Cmax of 1'-Hydroxymidazolam
Description: PK: Cmax of 1'-hydroxymidazolam
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug (midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.5 mg Midazolam | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20 | 20
ng/mL | 0.748 (40) | 0.722 (35)
Statistical Analysis 1: Comparison: 0.5 mg Midazolam vs 0.5 mg Midazolam + 400 mg Imlunestrant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; Ratio of Geometric least squares mean = 0.964, 90% CI 2-sided [0.828 to 1.12]

5. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to 24 Hours at Steady State (AUC[0-24], ss) of Imlunestrant When Dosed in the Presence of Midazolam
Description: PK: AUC[0-24], ss of Imlunestrant
Time Frame: Day 9: Predose, 0.25 h, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose
Population: All participants who received at least one dose of study drug (imlunestrant or midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20
ng*hr/mL | 2020 (53)

6. Secondary Outcome: PK: Maximum Observed Concentration at Steady State (Cmax, ss) of Imlunestrant When Dosed in the Presence of Midazolam
Description: PK: Cmax, ss of Imlunestrant when dosed in the presence of Midazolam is evaluated.
Time Frame: Day 9: Predose, 0.25 h, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h and 24h postdose
Population: All participants who received at least one dose of study drug (imlunestrant or midazolam) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.5 mg Midazolam + 400 mg Imlunestrant
Number analyzed (Participants) | 20
ng/mL | 120 (51)

ADVERSE EVENTS:
Time Frame: Baseline Up to Day 18
Description: All participants who received at least one dose of study drug (imlunestrant or midazolam). Participants were analyzed according to the treatment they actually received.
Groups:
- 400 mg Imlunestrant: Participants received 400 mg imlunestrant (2 × 200 mg) tablets administered QD orally for 7 days on Days 3 to 8.
Arm/Group | 0.5 mg Midazolam | 400 mg Imlunestrant | 0.5 mg Midazolam + 400 mg Imlunestrant
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 5/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg Midazolam (N=20) | 400 mg Imlunestrant (N=20) | 0.5 mg Midazolam + 400 mg Imlunestrant (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT05509816/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT05509816/SAP_001.pdf